CLINICAL TRIAL: NCT07018934
Title: Comparison of the Efficacy of Alpha-Blockers and Mirabegron on Symptoms Associated With Double-J Stent Implanted After Retrograde Intrarenal Surgery
Brief Title: Alfuzosin and Mirabegron for Double-J Stent Symptoms
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Mehmet Öztürk, Assoc. Prof., University of Gaziantep
Other Study IDs: 2024/05
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Ureteral Stent-Related Symptoms
Keywords: Nephrolithiasis; Ureteral Stent-Related Symptoms; Lower Urinary Tract Symptoms; Postoperative Pain; Retrograde Intrarenal Surgery
MeSH Terms: conditions — Nephrolithiasis; Lower Urinary Tract Symptoms; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Group 1 : The group that did not receive medical treatment
- 2: Group 2 : Alfuzosin 10 mg/d oral
- 3: Group 3 : Mirabegron 50 mg/d oral
- 4: Group 4 : Combination therapy with alfuzosin + Mirabegron

SUMMARY:
This prospective randomized controlled trial investigates the effects of alfuzosin, mirabegron, and their combination on stent-related symptoms and outcomes in patients undergoing DJ stent placement after retrograde intrarenal surgery (RIRS) for renal stones. The primary outcomes include stone-free rate and residual fragment status, while secondary outcomes focus on stent-related pain and lower urinary tract symptoms (LUTS). Patients will be randomly assigned to one of four groups: alfuzosin only, mirabegron only, combination therapy, or control. Pain and LUTS will be assessed using validated questionnaires such as the Ureteral Stent Symptom Questionnaire (USSQ) and IPSS.

DETAILED DESCRIPTION:
Retrograde intrarenal surgery (RIRS) is a commonly used minimally invasive procedure for the treatment of renal stones. Postoperative placement of double-J (DJ) stents is often necessary but can result in significant stent-related discomfort and lower urinary tract symptoms (LUTS), which negatively impact patient quality of life. Alfuzosin, an alpha-blocker, and mirabegron, a beta-3 agonist, are pharmacological agents known to reduce stent-related symptoms. This study aims to compare the individual and combined efficacy of these agents on stent-related pain, LUTS, and postoperative stone outcomes. Patients will be evaluated for stone clearance, residual fragments (by imaging), and symptom scores over a follow-up period of 2 to 4 weeks post-RIRS

ELIGIBILITY:
Inclusion Criteria:

- Undergoing RIRS and DJ stenting

Ability to provide informed consent

Exclusion Criteria:

* Neurogenic bladder

Prostate volume >40 mL or significant LUTS at baseline

Contraindications to alpha-blockers or mirabegron

Hepatic or severe renal impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 75 years undergoing retrograde intrarenal surgery (RIRS) for renal stones, followed by double-J (DJ) stent placement
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Stent-Related Pain Score | Day 7 postoperatively and Day 14 postoperatively.
  Pain score ranges from 0 to 39 (higher scores indicate worse pain).
Lower Urinary Tract Symptom (LUTS) Score | Day 7 postoperatively and Day 14 postoperatively
  IPSS ranges from 0 to 35 (higher scores indicate more severe LUTS).

SECONDARY OUTCOMES:
Stone-Free Rate | Day 14 postoperatively
  Proportion of patients with no residual fragments > 2 mm on NCCT
Residual Fragment Status | Day 14 postoperatively
  Categorization of residual fragments into 0 mm, 1-2 mm, or > 2 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University Faculty of Medicine Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to patient privacy concerns and institutional policy restrictions. However, summary results will be published in scientific journals and presented at academic meetings.

REFERENCES:
- [Result] Zhang K, Yan W, Li H, Chen J, Wang Q, Chai Y, Yuan L, Zhu G. Comparison of Mirabegron plus Tamsulosin and Tamsulosin Monotherapy for the Treatment of Ureteral Stent-Related Symptoms: A Prospective Randomized Study. Urol Int. 2022;106(12):1226-1232. doi: 10.1159/000526607. Epub 2022 Oct 14. PMID 36244331
- [Result] Uslu M, Yildirim U, Ezer M, Erihan IB, Sarica K. Residual fragment size following retrograde intrarenal surgery: a critical evaluation of related variables. Urolithiasis. 2023 Aug 9;51(1):100. doi: 10.1007/s00240-023-01478-8. PMID 37556003
- [Result] Geraghty RM, Davis NF, Tzelves L, Lombardo R, Yuan C, Thomas K, Petrik A, Neisius A, Turk C, Gambaro G, Skolarikos A, Somani BK. Best Practice in Interventional Management of Urolithiasis: An Update from the European Association of Urology Guidelines Panel for Urolithiasis 2022. Eur Urol Focus. 2023 Jan;9(1):199-208. doi: 10.1016/j.euf.2022.06.014. Epub 2022 Aug 1. PMID 35927160
- [Result] Yuk HD, Park J, Cho SY, Sung LH, Jeong CW. The effect of preoperative ureteral stenting in retrograde Intrarenal surgery: a multicenter, propensity score-matched study. BMC Urol. 2020 Sep 14;20(1):147. doi: 10.1186/s12894-020-00715-1. PMID 32928162

DOCUMENTS (1):
  • Study Protocol (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT07018934/Prot_000.pdf